CLINICAL TRIAL: NCT01785771
Title: An Open-Label Multi-Center Sub-Study to Evaluate the Efficacy, Safety and Tolerability of ITCA 650 in Patients With Type 2 Diabetes With High Baseline HbA1c
Brief Title: A Study to Evaluate ITCA 650 for the Treatment of Type 2 Diabetes in Patients With High Baseline HbA1c
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision by Sponsor
Sponsor: Intarcia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITCA 650-CLP-103-Sub-Study
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

ARMS (1):
- ITCA 650 (Experimental)
  Interventions: Drug: ITCA 650 (exenatide in DUROS)

INTERVENTIONS:
Drug: ITCA 650 (exenatide in DUROS)

SUMMARY:
An 39-week plus extensions, open-label study to estimate the reduction in HbA1c in patients with initial HbA1c >10% </=12% who are treated with ITCA 650 20 mcg/day for 13 weeks followed by ITCA 650 60 mcg/day for 26 weeks plus optional 26-week extensions with continued treatment with ITCA 650 60 mcg/day

ELIGIBILITY:
Inclusion Criteria:

* Men or women age 18 to 80 years with type 2 diabetes
* On stable treatment regimen of diet and exercise alone or in combination with a stable & optimal or near-optimal dose of metformin, sulfonylurea, TZD or combination of these drugs
* HbA1c >10.0% and ≤12.0%

Exclusion Criteria:

* Prior treatment with any GLP-1 receptor agonist
* History of hypersensitivity to exenatide or liraglutide
* FPG >300 mg/dL
* History of medullary thyroid cancer or a family or personal history of multiple endocrine neoplasia type 2
* Taking DPP-4 inhibitors, incretin mimetics, alpha glucosidase inhibitors, meglitinides or insulin within last 3 months
* history of pancreatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c between Week 39 and Day 0 | 39 weeks

CONTACTS AND LOCATIONS:
Locations (51):
- United States (51):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Fundamental Research, Gulf Shores, Alabama
  - East Valley Family Physicians, PLC, Chandler, Arizona
  - Desert Clinical Research, Mesa, Arizona
  - Clinical Research Advantage, Inc., Phoenix, Arizona
  - eStudySite, Chula Vista, California
  - Rocks Medical Research Institute, Inc., Fresno, California
  - Rocks Medical Research Institute, Fresno, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - Saviers Medical Group, Port Hueneme, California
  - University Clinical Investigatons, Inc/Diabetes Research Center, Tustin, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Colorado Springs Health Partners-Briargate, Colorado Springs, Colorado
  - Meridien Research, Bradenton, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - New Horizon Research Center, Inc., Miami, Florida
  - International Research Assocaites, LLC, Miami, Florida
  - Harmony Clinical Research, Inc., North Miami Beach, Florida
  - Palm Harbor Medical Associates, Palm Harbor, Florida
  - Andres Patron, D.O., P.A., Pembroke Pines, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Perimeter Institute for Clinical Research PRIME, Atlanta, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - Chicago Research Center, Chicago, Illinois
  - American Health Network of Indiana, LLC, Avon, Indiana
  - Medisphere Medical Research Center, LLC, Evansville, Indiana
  - American Health Network of Indiana, Franklin, Indiana
  - American Health Network of Indiana, LLC, Muncie, Indiana
  - Bunyan Clinical Research, Valparaiso, Indiana
  - Crescent City Clinical Research Center, Metairie, Louisiana
  - Palm Research Center, Inc., Las Vegas, Nevada
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - University of North Carolina at Chapel Hill, Durham, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Sentral Clinical Research Services, LLC, Cincinnati, Ohio
  - Columbus Clinical Research, Columbus, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Greer, South Carolina
  - BMG The Endocrine Clinic, Memphis, Tennessee
  - Tekton Research, Inc., Austin, Texas
  - 3rd Coast Research Associates, Corpus Christi, Texas
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Galena Research, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Medstar Clinical Research and Associates, Houston, Texas
  - Clinical Trials of Texas, Inc., San Angelo, Texas
  - Sound Healthcare, Port Orchard, Washington
  - Ranier Clinical Research Center, Renton, Washington

REFERENCES:
- [Derived] Henry RR, Rosenstock J, Denham DS, Prabhakar P, Kjems L, Baron MA. Clinical Impact of ITCA 650, a Novel Drug-Device GLP-1 Receptor Agonist, in Uncontrolled Type 2 Diabetes and Very High Baseline HbA1c: The FREEDOM-1 HBL (High Baseline) Study. Diabetes Care. 2018 Mar;41(3):613-619. doi: 10.2337/dc17-1519. Epub 2018 Jan 4. PMID 29301824